CLINICAL TRIAL: NCT01034176
Title: Effect of Fluoroquinolones on BK Viremia in the Renal Transplant Recipient, A Multi-Center Study
Brief Title: BK Treatment Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anil K. Chandraker, MD, Medical Director of Renal Transplantation, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009p000020
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: BK Viremia
Keywords: BK viremia; kidney transplantation; BK viremia in kidney transplant recipients
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levofloxacin (Active Comparator): Levofloxacin 500 mg every day (dose adjusted for renal function) for 30 days
  Interventions: Drug: levofloxacin
- placebo (Placebo Comparator): placebo identical to levofloxacin drug daily for 30 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levofloxacin — 500 mg tablet, daily, 30 days
  Other Names: Levaquin
  Arms: Levofloxacin
Drug: placebo — no dose, tablet, daily, 30 days
  Arms: placebo

SUMMARY:
Our hypothesis is that 30 days of oral levofloxacin (FDA approved antibiotic) in patients with persistent viremia (BK virus found in blood) will impair progress to BK virus induced kidney damage by significantly decreasing or eliminating BK virus in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Living and cadaveric kidney transplant recipients over the age of 18 years with BK viremia

Exclusion Criteria:

* Female patients of childbearing age who are pregnant or in whom adequate contraception cannot be maintained.
* Patients with active infections, history of malignancy/Posttransplant Lymphoproliferative Disease (PTLD) serologic positivity to HIV.
* Patients with evidence of urinary tract obstruction causing allograft dysfunction, unless corrected by time of enrollment.
* Patients with clinical or morphological evidence of recurrence of primary disease.
* Patients with a history of allergic reaction to quinolone antibiotics.
* Patients with history of prolong QT interval
* Patients with recurrent hypoglycemic episodes
* Patients with history of myasthenia gravis
* Patients taking Thioridazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chandraker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (8):
- United States (8):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Fletcher Allen Health Care/University of Vermont, Burlington, Vermont
  - University of Wisconsin Hospital, Madison, Wisconsin

REFERENCES:
- [Background] Leung AY, Chan MT, Yuen KY, Cheng VC, Chan KH, Wong CL, Liang R, Lie AK, Kwong YL. Ciprofloxacin decreased polyoma BK virus load in patients who underwent allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2005 Feb 15;40(4):528-37. doi: 10.1086/427291. Epub 2005 Jan 21. PMID 15712075
- [Background] Randhawa PS. Anti-BK virus activity of ciprofloxacin and related antibiotics. Clin Infect Dis. 2005 Nov 1;41(9):1366-7; author reply 1367. doi: 10.1086/497080. No abstract available. PMID 16206122
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Lee BT, Gabardi S, Grafals M, Hofmann RM, Akalin E, Aljanabi A, Mandelbrot DA, Adey DB, Heher E, Fan PY, Conte S, Dyer-Ward C, Chandraker A. Efficacy of levofloxacin in the treatment of BK viremia: a multicenter, double-blinded, randomized, placebo-controlled trial. Clin J Am Soc Nephrol. 2014 Mar;9(3):583-9. doi: 10.2215/CJN.04230413. Epub 2014 Jan 30. PMID 24482066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levofloxacin | Placebo
Started | 22 | 21
Completed | 20 | 19
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Full Range); unit: years] — Age at time of consent
  years
    Age at time of consent | 56.22 [32 to 74] | 54.9 [25 to 70] | 55.36 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in BK Virus Copies at 3 Months
Description: Percent change in BK virus copies/mL from Baseline to 3 months
Time Frame: Baseline and 3 months
Measure: Median (Standard Deviation); unit: Percent change of BK virus copies
Arm/Group | Levofloxacin | Placebo
Number analyzed (Participants) | 20 | 19
Percent change of BK virus copies | 70.3 (42.5) | 69.1 (39.5)

2. Secondary Outcome: Number of Patients With >50% Reduction in BK Virus Copies
Description: Number of patients with >50% reduction in BK viral load at 6 months
Time Frame: Baseline and 6 months
Population: number of patients with >50% reduction in BK viral load at 6 months
Measure: Number; unit: participants
Arm/Group | Levofloxacin | Placebo
Number analyzed (Participants) | 20 | 19
participants | 15 | 13

ADVERSE EVENTS:
Arm/Group | Levofloxacin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/19
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/19
Other Adverse Events (participants affected / at risk) | 2/20 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=20) | Placebo (N=19)
Neoplasm, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — unrelated
suicidal ideation (Psychiatric disorders) | 0 | 1 — unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=20) | Placebo (N=19)
achilles tendon strain/injury (Musculoskeletal and connective tissue disorders) | 2 | 0 — possibly related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No